CLINICAL TRIAL: NCT01691209
Title: An Investigator-blinded, Randomized, Monocentre, 3-arm, Active Controlled Pilot Trial to Explore the Efficacy and Safety of a Topical Medical Device in Patients With Mild to Moderate Atopic Dermatitis in an Intra-individual Comparison With a Standard Therapy (1% Hydrocortisone Cream) and Untreated Skin
Brief Title: Efficacy/Safety Study to Explore a New Topical Formulation in Atopic Dermatitis
Acronym: Phoenix
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Head Medical Affairs, Bayer HealthCare AG, Consumer Care
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16200; 2012-001504-38 (EudraCT Number)
Record Dates: First submitted 2012-09-20; First posted 2012-09-24 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Dermatitis, Atopic
Keywords: Phoenix; Hydrocortison; mild atopic dermatitis; efficacy; safety
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Phoenix (Experimental): Application over 29 days twice daily
  Interventions: Device: Phoenix (BAY81-2996)
- Hydrocortison (Active Comparator): Application over 29 days twice daily
  Interventions: Drug: 1% Hydrocortison cream
- Untreated skin (No Intervention): Participants will be observed over 29 days without study treatment

INTERVENTIONS:
Device: Phoenix (BAY81-2996) — Topical formulation applied to the skin
  Arms: Phoenix
Drug: 1% Hydrocortison cream — 1% Hydrocortison cream applied to the skin
  Arms: Hydrocortison

SUMMARY:
The study shall explore whether treatment of atopic dermatitis is equally effective with Phoenix medical device as compared to standard therapy (Hydrocortisone cream).

ELIGIBILITY:
Inclusion Criteria:

* Male or female Caucasians aged between 18 and 60 years
* Patients with mild atopic dermatitis (AD) presenting a scoring AD (SCORAD) rating below 50
* Skin type I - IV according to Fitzpatrick
* Acute AD symptoms on each assessment areas (local SCORAD ≥ 3 and <= 12) at Baseline
* Acute symptom of pruritus at Baseline

Exclusion Criteria:

* Any other skin disease at the test area that would interfere with the clinical assessment in the opinion of the investigator
* Moles, tattoos, strong pigmentation, or scars at the test area that would interfere with the clinical assessment
* Regular intake of antiphlogistic drugs (for example nonsteroidal anti-inflammatory drugs [NSAIDs])
* Any condition or treatment which might influence the trial (e.g. any treatment with topical antibiotics, antifungals, or corticoids) within 14 days prior to screening as well as during the trial (exception: topical treatment of AD lesions other than the test areas (for example, face) with low potency steroids restricted to small areas)
* UV-therapy or the use of solarium within 30 days before screening as well as during the trial
* Any alternative treatment of AD (e.g. acupuncture, kinesiology, and homoeopathy) within 30 days before screening as well as during the trial

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2014-04 (Estimated); Study Completion 2014-06 (Estimated)

SECONDARY OUTCOMES:
Number of participants with abnormal vital signs | Up to 10 weeks
  Vital signs consist of blood pressure, heart rate and body temperature.
Number of participants with adverse events as a measure of safety and tolerability | Up to 10 weeks

OTHER OUTCOMES:
Local scored atopic dermatitis (SCORAD) as clinical assessment by means of the intensity items of the SCORAD index | Up to 29 days
Transepidermal water loss (TEWL) as a measure for skin barrier function | Up to 29 days
Skin hydration by means of corneometry | Up to 29 days
Erythema by means of chromametry | Up to 29 days
Intensity of pruritus by means of visual analogue scale (VAS) | Up to 29 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Münster, North Rhine-Westphalia, Germany